CLINICAL TRIAL: NCT01904552
Title: Influence of Apical Periodontitis on the Accuracy of Three Electronic Root Canal Length Measurement Devices: An In Vivo Study
Brief Title: Accuracy of ERCLMDs in Teeth With Apical Periodontitis
Acronym: ERCLMDs
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Isfahan University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Masoud Saatchi, Isfahan University of Medical Sciences, Isfahan University of Medical Sciences
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Grant: 390553; Grant: 390553 (Other: Isfahan University of Medical Sciences); 39232 (Other: Isfahan University of Medical Sciences)
Record Dates: First submitted 2013-07-11; First posted 2013-07-22 (Estimated); Last update posted 2013-07-22 (Estimated); Status verified 2013-07

CONDITIONS: Apical Periodontitis
Keywords: Apical periodontitis; Dentaport ZX; electronic apex locators; i-Root; Raypex 5; working length
MeSH Terms: conditions — Periapical Periodontitis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- apical periodontitis (AP) (Experimental): clinical pulp necrosis periapical index scores of 3, 4 or 5
  Interventions: Device: Electronic Root Canal Length Measurement Device
- normal periapex (NP) (Experimental): clinical pulp vitality periapical index score of 1
  Interventions: Device: Electronic Root Canal Length Measurement Device

INTERVENTIONS:
Device: Electronic Root Canal Length Measurement Device — Electronic Apex Locator is used to find the apical foramen of the root canal. It uses a weak electrical current passed through the canal by endodontic file
  Other Names: Dentaport ZX; Raypex; i-Root

SUMMARY:
The aim of this in vivo study is to evaluate the influence of apical periodontitis (AP) on the accuracy of Dentaport ZX, Raypex 5, and i-Root electronic root canal length measurement devices.

DETAILED DESCRIPTION:
Thirty-two single-rooted teeth scheduled for extraction, consisting of 16 teeth with AP and 16 teeth with normal periapex (NP), were selected. Access cavity was prepared and coronal portion of the canal was flared. Electronic working length (EWL) was determined by each ERCLMD according to each manufacturer's instructions. Each tooth was extracted and actual working length (AWL) was determined by inserting a size 15 K-file until the tip could be seen at a position tangential to the major foramen and then 0.5 mm was subtracted from the measurement. The distance from the AWL to the file tip was calculated and compared between the two groups by t-test. The accuracy of each ERCLMD within ±0.5 mm was compared between the groups by Fisher's test. Statistical significance was set at P < .05.

ELIGIBILITY:
Inclusion Criteria:

* single-rooted teeth
* clinical pulp necrosis and periapical index scores of 3, 4 or 5
* pulp vitality and a periapical index score of 1

Exclusion Criteria:

* Teeth with metal restorations
* Teeth with prosthetic crowns
* Teeth with pulp calcification
* Teeth with previous endodontic treatment

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2012-09; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Actual working length (AWL) | 6 months

SECONDARY OUTCOMES:
Electronic working length (EWL) | 6 months

OTHER OUTCOMES:
working length | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Masoud Saatchi, DDS MS, Principal Investigator — Isfahan University of Medical Sciences
Locations (1):
- Isfahan University of Medical Sciences, Isfahan, Isfahan, Iran

REFERENCES:
- See also: Isfahan University of Medical Sciences — http://mui.ac.ir/en/